CLINICAL TRIAL: NCT01352936
Title: Comparison of Nephrotoxicity and Hospital Costs in Patients With Methicillin-Resistant Staphylococcus Aureus Bacteremia Who Received Vancomycin Versus Teicoplanin Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yuh-Mou Sue, Department of Internal Medicine, Wanfang Hospital
Other Study IDs: 100007
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Staphylococcus Aureus; Bacteremia
Keywords: nephrotoxicity; hospital cost; Staphylococcus aureus; bacteremia; vancomycin; teicoplanin
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
Staphylococcus aureus, the most virulent of the many staphylococcal species, has been recognized as one of the most important and lethal human bacterial pathogens. With the increased incidence of methicillin-resistant staphylococcus aureus (MRSA) infection in community and hospitalized patients, MRSA infections are associated with greater lengths of stay, higher mortality, and increased costs. Vancomycin and teicoplanin, are the two most commonly used glycopeptides and are the first-choice of treatment for MRSA infection. Vancomycin-induced nephrotoxicity is still a point of controversy. Teicoplanin is not known to have any nephrotoxicity. Acute kidney injury is a common complication of critical illness, which is reported in 5 to 7% of hospitalized patients. It is associated with significantly increased mortality, length of stay, and costs across a broad spectrum of conditions.

DETAILED DESCRIPTION:
In this retrospective observational study, data collection was performed using the patient list extracted from the medical management system of Taipei Medical University-Wan Fang Hospital. Hospitalized patients who had been prescribed either vancomycin or teicoplanin for treating bloodstream infection caused by MRSA and had at least one serum creatinine data within 7 days after initiating glycopeptide therapy were recruited for this study. The major outcome variables of interest were the new onset of nephrotoxicity, which was defined as decrease of glomerular filtration rate (GFR) for more than 25% or 50% from baseline based on serial serum creatinine (SCr) measurements. Other variables including age at admission, gender, comorbidities, laboratory data, concurrent medications (e.g., drug name, dose, route, dosing interval, starting date and end date), and medical cost information were also obtained from the database.

We performed this observational clinical study with 2 main goals: (1) to determine the rate of nephrotoxicity and mortality in patients with MRSA bacteremia treated with vancomycin or teicoplanin; (2) to determine whether vancomycin-associated nephrotoxicity increase length of stay and costs.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who had been prescribed either vancomycin or teicoplanin for treating bloodstream infection caused by MRSA and had at least one serum creatinine data within 7 days after initiating glycopeptide therapy were recruited for this study.

Exclusion Criteria:

* Patients who aged less than 15 years at admission were excluded. Those who switch treatment from vancomycin to teicoplanin or vise versa during the hospitalization were also excluded to avoid any possible carryover effect. Because the main objectives of this study were to compare the magnitude and consequences of nephrotoxicity associated with the two study medications, patients who underwent dialysis before the glycopeptides treatment were further excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Staphylococcus aureus patients
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2011-01; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Mou Sue, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan